CLINICAL TRIAL: NCT06184646
Title: Effect of Calcium and Vitamin D Supplements and/or Prunes on Bone Health
Brief Title: Elucidating the Minimal Effective Dose of Prunes for Bone Health in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Shirin Hooshmand, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-2023-0243
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Bone Disease, Metabolic
Keywords: Osteopenia; Prune; Functional food
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (0 g prune/day) (No Intervention): Participants only receive 500 mg calcium and 400 IU vitamin D daily for 24 months.
- 30 g prune/day (Experimental): Participants receive 500 mg calcium and 400 IU vitamin D daily for 24 months and 30 g of prune daily for 24 months.
  Interventions: Dietary Supplement: Prune

INTERVENTIONS:
Dietary Supplement: Prune — 30 g of prune/day
  Arms: 30 g prune/day

SUMMARY:
The objective of this study is to examine if calcium and vitamin D supplements and/or prune can prevent bone loss in postmenopausal women.

DETAILED DESCRIPTION:
Two hundred randomly assigned to one of two treatment groups: 1) 30 g prunes and 2) control (0 g prunes). Both groups received 500 mg calcium and 400 IU Vitamin D as a daily supplement. Blood samples are collected at baseline, 12 and 24 months to assess biomarkers of bone turnover. Physical activity recall and food records are obtained at baseline, 12 and 24 months to examine physical activity and dietary confounders as potential covariates. Dual-energy x-ray absorptiometry (DXA) and peripheral quantitative computed tomography (pQCT) will be completed at baseline, 12 and 24 months to examine bone mineral density and structure.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* BMD t-score is between 0.5 and 2 SD below the mean
* Not on hormone replacement therapy (HRT) and/or other pharmacological agents known to affect bone for at least three months prior to initiation of the study

Exclusion Criteria:

* Women whose BMD t-score at any site falls below 2.5 SD of the mean
* Subjects receiving endocrine (e.g., prednisone, other glucocorticoids) or neuroactive (e.g., dilantin, phenobarbital) drugs or any drugs known to influence bone and calcium metabolism
* Subjects who smoke cigarettes or vape
* Regular consumption of dried plum or prune juice

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in bone mineral density at 12 and 24 months | Baseline, 12 months, and 24 months
  bone mineral density as assessed by dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Changes from baseline in bone specific alkaline phosphatase at 12 months and 24 months | Baseline, 12 months, and 24 months
  bone specific alkaline phosphatase (BAP) as assessed with ELISA
Changes from baseline in tartrate acid phosphatase-5b at 12 months and 24 months | Baseline, 12 months, and 24 months
  tartrate acid phosphatase-5b (TRAP5b) as assessed with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No